CLINICAL TRIAL: NCT07009639
Title: Evaluation of Artificial Intelligence-Assisted Echocardiography (AI-echo) in the Early Diagnosis and Prognostic Stratification of Left Atrial Cardiomyopathy (LACM) in Patients With Acute Cardiac Disease
Brief Title: Prognostic Role of AI-Echo
Status: Recruiting | Type: Observational
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Antonio Curcio, Professor, University of Calabria
Other Study IDs: 58/2025
Record Dates: First submitted 2025-05-15; First posted 2025-06-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Atrial Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Left atrial cardiomyopathy (LACM) is frequently underdiagnosed but plays a key role in increasing the risk of atrial fibrillation (AF) and thromboembolic events. While atrial strain is a validated marker of LACM, its measurement with conventional echocardiography can be time-consuming and less feasible in acute settings. The use of AI-assisted echocardiography (AI-echo) may help streamline image acquisition and analysis, offering faster and potentially more accurate assessment.

This study aims to compare the time required for atrial strain analysis using AI-echo versus standard methods. It also explores how changes in strain parameters (LASr, LASct, LAScd) relate to the onset of AF and in-hospital adverse outcomes, adjusting for comorbidities and conventional echo variables.

Main endpoints include time reduction with AI-echo and the association between strain changes and AF, complications, or mortality during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Hospitalization in CCU for acute cardiac pathology (e.g. acute coronary syndrome, acute or exacerbated heart failure, malignant arrhythmias, etc.).
3. Ability to provide written informed consent.

Exclusion Criteria:

1. Severe hemodynamic instability, history to contraindicate the execution of the echocardiographic examination.
2. Severely inadequate echocardiographic window that precludes atrial or ventricular morpho-functional assessment.
3. Inability to continue the study for clinical reasons, logistics or patient refusal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-85 years, in sinus rhythm at the time of enrollment, with an indication for echocardiography for acute cardiac pathology.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic acquisition times changes | From the start of echocardiographic acquisition to the completion of atrial strain analysis
  To compare the duration of echocardiographic image acquisition and atrial strain analysis using an AI-assisted echocardiography software versus the conventional manual method in patients admitted to the Cardiac Intensive Care Unit (CCU). All measurements will be performed using the same ecocardiography machine and by the same operator to ensure consistency. The outcome will be assessed by measuring the time (in minutes) required to complete image acquisition and atrial strain analysis with each method.
Change in left atrial reservoir strain (LASr) between admission and discharge | At admission (within 24 hours of enrollment) and at discharge (within 24 hours before discharge)
  To assess the variation in left atrial reservoir strain (LASr), measured by speckle-tracking echocardiography, between hospital admission and discharge in patients admitted to the Cardiac Intensive Care Unit (CCU). Measurements will be performed in each patient at two time points: within 24 hours of admission and within 24 hours prior to discharge.
Change in left atrial conduit strain (LAScd) between admission and discharge | At admission (within 24 hours of enrollment) and at discharge (within 24 hours before discharge)
  To assess the variation in left atrial conduit strain (LAScd), measured by speckle-tracking echocardiography, between hospital admission and discharge in patients admitted to the Cardiac Intensive Care Unit (CCU). Measurements will be performed in each patient at two time points: within 24 hours of admission and within 24 hours prior to discharge.
Change in left atrial contractile strain (LASct) between admission and discharge Description | At admission (within 24 hours of enrollment) and at discharge (within 24 hours before discharge)
  To assess the variation in left atrial contractile strain (LASct), measured by speckle-tracking echocardiography, between hospital admission and discharge in patients admitted to the Cardiac Intensive Care Unit (CCU). Measurements will be performed in each patient at two time points: within 24 hours of admission and within 24 hours prior to discharge.
Correlation between atrial strain variation (ΔLASr, ΔLASct, ΔLAScd) and in-hospital heart failure worsening | From admission (within 24 hours of enrollment) to discharge (within 24 hours before discharge)
  To evaluate whether changes in atrial strain parameters (ΔLASr, ΔLASct, ΔLAScd), measured via speckle-tracking echocardiography, correlate with the incidence of in-hospital worsening of heart failure (Unit of Measure: % of patients with in-hospital worsening heart failure). Worsening is defined as the need for intensification of diuretic therapy, initiation of inotropes, transfer to higher-level care, or an increase in NT-proBNP levels compared to baseline (measured in pg/mL).

SECONDARY OUTCOMES:
Incidence of in-hospital procedural complications | Through study completion, an average of 7 days
  To assess the incidence of complications (% of patients with at least one procedural complication) related to diagnostic or interventional procedures during hospitalization, including but not limited to pericardial effusion, vascular access complications, and device-related issues. Events will be recorded based on clinical documentation and adjudicated by the clinical team.
Incidence of in-hospital infections | Through study completion, an average of 7 days
  To assess the incidence of infections acquired during hospitalization (% of patients with at least one in-hospital infection), defined by clinical diagnosis supported by laboratory/microbiological findings and initiation of antimicrobial therapy.
Incidence of in-hospital thromboembolic events | Through study completion, an average of 7 days
  To assess the incidence of thromboembolic events (% of patients with at least one thromboembolic event) during hospitalization, including ischemic stroke, systemic embolism, deep vein thrombosis, or pulmonary embolism, confirmed by imaging and/or laboratory criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- "Annunziata" Hospital, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No